CLINICAL TRIAL: NCT05955391
Title: A Multi-centered, Open-label, Single-arm Phase II Study to Evaluate the Safety and Efficacy of TGRX-326 Monotherapy in Patients of Advanced ALK-positiveNon-Small Cell Lung Cancer Who Failed 2nd-Generation ALK Inhibitor Therapies
Brief Title: TGRX-326 Chinese Phase II for Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Sun Yat-sen University (Other); Tongji Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); The First Affiliated Hospital of Zhengzhou University (Other); West China Hospital (Other); Zhejiang University (Other); Jilin Provincial Tumor Hospital (Other); Hunan Cancer Hospital (Other); Shandong Cancer Hospital and Institute (Other); Jiangxi Provincial Cancer Hospital (Other); First Hospital of China Medical University (Other); The Affiliated Hospital of Qingdao University (Other); Liaoning Cancer Hospital & Institute (Other); Haerbin Medical University Cancer Hospital (Unknown); Xinxiang Central Hospital (Other); Xiangyang Central Hospital (Other); Mianyang Central Hospital (Other); Zhejiang Cancer Hospital (Other); Henan Cancer Hospital (Other Government); First Affiliated Hospital, Sun Yat-Sen University (Other); First Affiliated Hospital of Bengbu Medical College (Unknown); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Bingzhou Medical University Affiliated Hospital (Unknown); Fujian Cancer Hospital (Other Government); Ningbo No. 1 Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Second Affiliated Hospital of AFMU (Unknown); Yunnan Cancer Hospital (Other); Capital Medical School Beijing Chest Hospital (Unknown); Shijiazhuang People's Hospital (Other); Tianjin Cancer Hospital (Unknown); Affiliated Cancer Hospital of Guizhou Medical University (Unknown); Nanchang University First Affiliated Hospital (Unknown); Jingzhou First People's Hospital (Unknown); Shanghai Chest Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-326-2001-NSCLC-CN
Record Dates: First submitted 2023-07-10; First posted 2023-07-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: TGRX-326 (Experimental): Subjects to be treated with the investigational drug TGRX-326 at 60 mg once day in 21-day cycles.
  Interventions: Drug: TGRX-326

INTERVENTIONS:
Drug: TGRX-326 — Subjects will be treated with the investigational drug TGRX-326 at 60 mg once day in 21-day cycles

SUMMARY:
This is a multi-center, single-arm, open-label, Phase II clinical trial which explores the safety and efficacy of TGRX-326 in patients with ALK-positive advanced NSCLC who have failed prior 2nd-generation ALK treatments due to progressive disease or intolerance.

DETAILED DESCRIPTION:
This Phase II studyaims to evaluate the safety profile and efficacy profile in patients with ALK-positive advanced NSCLC. The primary purpose of this study is to evaluate the efficacy profile of TGRX-326, with the objective response rate (ORR) as end point. Secondary objectives include evaluating efficacy profile of other endpoints and safety profiles of the investigational drug. Exploratory objective includes the evaluation of population pharmacokinetic (PK) profile of TGRX-326.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to follow the treatment protocol and visit schedule, and participate in the study with the ICF signed;
2. ≥ 18 years of age on the day of ICF signing, regardless of gender.
3. With ALK-positive advanced inoperable NSCLC and having disease progression or intolerance after continuous treatment with second-generation ALK inhibitors;
4. Providing prior ALK positive test results at screening;
5. Patients could have metastases to central nervous system at screening if the condition is asymptomatic, stable or completely recovered;
6. Drug discontinuation for ≥ 5 half-lives prior to the first dose for subjects previously treated with ALK inhibitors;
7. At least one measurable lesion;
8. An ECOG PS score within 0-2;
9. Adequate bone marrow, liver, kidney, coagulation and pancreatic functions;
10. Expected survival ≥ 3 months;
11. Willing to take effective contraceptive measures (for men of reproductive potential and women of reproductive age only) from ICF signing to 6 months after administration of the investigational drug. Women of reproductive age include women before menopause and within 2 years after menopause. Those women must have a negative pregnancy test ≤ 7 days prior to the first dose of the investigational drug.

Exclusion Criteria:

1. Previous use of any third-generation ALK inhibitors other than TGRX-326;
2. Known hypersensitivity to any of the active ingredients or excipients of TGRX-326 or a history of severe allergic reactions that makes himself/herself unsuitable for TGRX-326 treatment in the judgment of the investigator;
3. Having another type of cancer except for lung cancer;
4. Major surgery within 4 weeks prior to the first dose;
5. Spinal cord compression caused by tumor, unless the subject achieves significant pain control and full recovery of neurological function within 4 weeks prior to the first dose.
6. Abnormal gastrointestinal function that affect absorption within the past 6 months;
7. History of active pneumonia or clinically significant interstitial pneumonia, or radiation or drug-induced lung disorder with treatment needs;
8. Cardiac insufficiency;
9. Abnormal and clinically significant QTc on ECG or need of concomitant use of any drug known to prolong QT interval and cause torsades de pointes;
10. Uncontrolled hypertension after drug treatment;
11. Uncontrolled hyperglycaemia, acute attack of cholelithiasis, and susceptibility to acute pancreatitis;
12. Severe or uncontrolled systemic diseases causing expected intolerance to the investigational drug as judged by the investigator;
13. Use within 14 days before the first dose or expected concomitant use during the treatment period of drugs that pose risk of QTC interval prolongation and/or ventricular tachycardia;
14. Previous antineoplastic treatments within 28 days prior to the first dose of the investigational drug;
15. Toxic reactions associated with prior surgery and prior antineoplastic therapies that have not recovered and may affect the subject safety as assessed by the investigator.
16. Clinically significant active bacterial, fungal or viral infections, including a positive result for hepatitis B surface antigen and HBV DNA ≥ ULN, one or more positive results for hepatitis C antibody or HIV antibody, or the presence of any uncontrolled infection.
17. Use of strong CYP3A4 inducers or inhibitors or CYP3A4 substrates with a narrow therapeutic window within two weeks prior to the first dose of the investigational drug;
18. Pregnant and breastfeeding female;
19. Women of childbearing age who are unwilling or unable to use acceptable methods for contraception during the entire treatment period in the trial and within 6 months after the last dose of the investigational drug (women of childbearing age include: any one with menarche, and those who have not received successful artificial sterilization [hysterectomy, bilateral fallopian tube ligation, or bilateral oophorectomy] or premenopausal women); a fertile male patient who is unwilling or unable to take effective contraceptive measures, and whose partner is a woman of childbearing age;
20. Being involved in other clinical studies (except for the non-interventional phase of interventional clinical study, such as survival follow-up period); less than 4 weeks from the end of the dose of other investigational drug to the first dose of the investigational drug or 5 half-lives of the previous drug, whichever is shorter;
21. Any mental or cognitive disorders which may limit subjects' understanding and implementation of the informed consent form;
22. Other situations, such as poor compliance, which are considered by the investigator to be not suitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  ORR defined by the ratio of patients who reachedthe treatment response; ORR as evaluated by independed review committee (IRC)

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  DCR defined by the ratio of patients who reached the treatment response or maintained as stable desease; DCR as evaluated by IRC and investigator
Duration of Response (DOR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  DOR defined as the duration from first occurence of treatment response to progressive disease/relapse; DOR as evaluated by IRC and investigator
Time to Response (TTR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  TTR defined by the time from the start of treatment to the first ORR; TTR as evaluated by IRC and investigator
Progression Free Survival (PFS) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  PFS defined by the time from randomization to progressive disease or death of any cause; PFS as evaluated by IRC and investigator.
Intracranial Objective Response Rate (IC-ORR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  IC-ORR defined by the ratio of patients who reached the intracranial treatment response; ORR as evaluated by independed review committee (IRC) and investigator.
Intracranial Disease Control Rate (IC-DCR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  IC-DCR defined by the ratio of patients who reached the treatment response intracranially or maintained as stable desease; IC-DCR as evaluated by IRC and investigator
Intracranial Duration of Response (IC-DOR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  IC-DOR defined as the duration from first occurence of Intracranial treatment response to progressive disease/relapse; DOR as evaluated by IRC and investigator
Intracranial Time to Response (IC-TTR) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  IC-TTR defined by the time from the start of treatment to the first IC-ORR; TTR as evaluated by IRC and investigator
Intracranial Progression Free Survival (IC-PFS) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  IC-PFS defined by the time from randomization to progressive disease or death of any cause inpatients with intracranial lesions; PFS as evaluated by IRC and investigator.
Overall Survival (OS) | Every 2 cycles between Cycle 1 and Cycle 17, and every 12 weeks from Cycle 17 and onwards (every cycle is 21 days); an average of 1.5 years
  OS defined by the time from randomization to death of any cause; PFS as evaluated by IRC and investigator.
Adverse Events (AEs) | Through completion of the study, an average of 1.5 years
  To record and analyse subjects with adverse events (AEs)
Serious Adverse Events (SAEs) | Through completion of the study, an average of 1.5 years
  To record and analyse subjects with serious adverse events (SAEs)

OTHER OUTCOMES:
Plasma Cmax | Day 1 of Cycle 1, 3, 5, 7, and every 2 cycles until cycle 17 (each cycle is 21 days)
  Cmax of TGRX-326 as measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Study Principal Investigator
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No